CLINICAL TRIAL: NCT02716012
Title: A First-in-Human, Multi-centre, Open-label, Phase 1a/b Clinical Study With RNA Oligonucleotide Drug MTL-CEBPA to Investigate Its Safety, Tolerability, and Antitumour Activity in Patients With Advanced Liver Cancer
Brief Title: First-in-Human Safety, Tolerability and Antitumour Activity Study of MTL-CEBPA in Patients With Advanced Liver Cancer
Acronym: OUTREACH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mina Alpha Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNA-3521-011; 2015-003051-21 (EudraCT Number); 20332 (Other: UK NIHR CRN)
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Oligonucleotide; RNA; saRNA; Sorafenib; Myeloid
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MTL-CEBPA Monotherapy (Experimental): MTL-CEBPA administered weekly, twice weekly or thrice weekly over 3 weeks followed by 1 week of rest defining a 28-day cycle.
  Interventions: Drug: MTL-CEBPA
- MTL-CEBPA & Sorafenib (combination) (Experimental): MTL-CEBPA is administered weekly or twice weekly in combination with sorafenib over 3 weeks followed by 1 week of rest defining a 28-day cycle.
  Interventions: Drug: MTL-CEBPA; Drug: Sorafenib 200mg
- MTL-CEBPA & Sorafenib (sequential) (Experimental): MTL-CEBPA is administered weekly or twice weekly for 2 cycles (28-day cycle) followed by 2 cycles of sorafenib
  Interventions: Drug: MTL-CEBPA; Drug: Sorafenib 200mg

INTERVENTIONS:
Drug: MTL-CEBPA — Intravenous administration
Drug: Sorafenib 200mg — Sorafenib tablets
  Arms: MTL-CEBPA & Sorafenib (combination); MTL-CEBPA & Sorafenib (sequential)

SUMMARY:
MNA-3521-011 study is a multi-centre, open-label, first-in-human, phase 1a/b clinical study dose/dose frequency escalation followed by a cohort expansion part. MTL-CEBPA is administered as monotherapy or in combination with sorafenib to patients with advanced hepatocellular carcinoma and cirrhosis of the liver. All participants will be considered unsuitable for liver tumour resection and/or is refractory to radiotherapy and other loco-regional therapies.

MTL-CEBPA consists of a double stranded RNA formulated into a SMARTICLES® liposomal nanoparticle and is designed to activate the CEBPA gene.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced HCC with cirrhosis resulting from hepatitis B, hepatitis C, alcohol-related liver disease or any other aetiology OR Histologically confirmed advanced HCC resulting from NASH with or without cirrhosis
* Patient is considered unsuitable for liver tumour resection and/or is refractory to radiotherapy and other loco-regional therapies
* At least one measurable lesion with target lesion size ≥ 1.0 cm as measured by MRI or CT
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Child-Pugh class A or B (up to B7)
* Eligible to undergo pre and post treatment mandated biopsies
* Acceptable laboratory parameters, as demonstrated by:

  * Platelets ≥ 70 x 10^9/L
  * Serum albumin > 26 g/L
  * ALT and AST ≤ 5 x ULN
  * Bilirubin ≤ 50 µmol /L
  * WBC ≥ 2.0 x 10^9/L, Absolute neutrophil count ≥ 1.5 x 109/L
  * Haemoglobin ≥ 9.0 g/dL
  * Prothrombin time (PT) <20 seconds
* Acceptable renal function as demonstrated by:

  * Serum creatinine ≤ 1.5 x ULN
  * Calculated creatinine clearance ≥ 60 mL/min

Exclusion Criteria:

* Patients who have been treated with TACE or chemotherapy within the last 28 days
* Prior investigational drugs within the last 30 days
* Grade > 1 prior treatment-related toxicities (excluding alopecia) at the time of screening
* Patients with clinically significant cancer ascites
* Any episode of bleeding from oesophageal varices or other uncontrolled bleeding within the last 3 months prior to study treatment initiation
* Patients with history of haemorrhage or gastrointestinal perforation
* Patients administered with serum albumin within the last 7 days prior to the first study drug administration
* Known infection with human immunodeficiency virus (HIV)
* Patients with central nervous system (CNS), bone or peritoneal metastasis
* Patients presenting with marked baseline prolongation of QT/QTc interval defined as repeated demonstration of a QTc interval ≥450 ms (males) and ≥460 ms (females) using Fridericia's correction formula
* Signs and symptoms of heart failure characterised as greater than the New York Heart Association (NYHA) Class I or other clinically significant cardiac abnormalities (including history of myocardial infarction) including stable abnormalities.
* Major surgery within the last 30 days prior to study treatment initiation
* Patients with history of organ transplantation or cardiac surgery
* Patients with sepsis, ineffective biliary drainage with or without cholangitis, obstructive jaundice or encephalopathy at screening visit or within the last two weeks prior to study treatment initiation, whichever earlier
* Evidence of spontaneous bacterial peritonitis or renal failure or allergic reactions to the agent or excipient at screening visit or within the last two weeks prior to study treatment initiation, whichever earlier
* Known hypersensitivity to the active sorafenib or to any of the excipients
* Occurrence of a grade 3 or higher sorafenib or lenvatinib related toxicity during any sorafenib / lenvatinib treatment received prior to study enrolment, according to toxicity criteria (NCI CTCAE v 5.0)
* Pregnant or lactating women

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1- Incidence of Grade 3 or 4 drug related adverse events | During cycle 1 (28 days) of treatment assessed over 15 months
  Frequency of adverse events graded according to NCI CTCAE v5.0
Part 2 - Change in tumour size from baseline using RECIST 1.1 and mRECIST in patients treated with MTL-CEBPA in combination with sorafenib | Eight weekly intervals until death assessed for 100 weeks
  Increase or decrease in tumour measurement using Response Evaluation Criteria in Solid Tumours (RECIST) reports

SECONDARY OUTCOMES:
Part 2 - Safety and tolerability of co-administering MTL-CEBPA with sorafenib assessed using frequency of adverse events graded according to toxicity criteria (NCI CTCAE v 5.0) and categorised by body system | At the end of every cycle (28 days) of treatment assessed over 15 months
  Frequency of treatment-related adverse events graded according to NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dr Debashis Sarker, MBChB, MRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust and King's College London; Professor Nagy Habib, FRCS, Study Director — Mina Alpha Limited
Locations (11):
- National University Hospital, Singapore, Singapore
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (9):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Trust, Cambridge
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Royal Free London NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarker D, Plummer R, Meyer T, Sodergren MH, Basu B, Chee CE, Huang KW, Palmer DH, Ma YT, Evans TRJ, Spalding DRC, Pai M, Sharma R, Pinato DJ, Spicer J, Hunter S, Kwatra V, Nicholls JP, Collin D, Nutbrown R, Glenny H, Fairbairn S, Reebye V, Voutila J, Dorman S, Andrikakou P, Lloyd P, Felstead S, Vasara J, Habib R, Wood C, Saetrom P, Huber HE, Blakey DC, Rossi JJ, Habib N. MTL-CEBPA, a Small Activating RNA Therapeutic Upregulating C/EBP-alpha, in Patients with Advanced Liver Cancer: A First-in-Human, Multicenter, Open-Label, Phase I Trial. Clin Cancer Res. 2020 Aug 1;26(15):3936-3946. doi: 10.1158/1078-0432.CCR-20-0414. Epub 2020 May 1. PMID 32357963
- See also: Company Webpage — http://minatx.com